CLINICAL TRIAL: NCT04446546
Title: Long Term Outcomes of Cold Stored Venous Allografts in Vascular Access for Hemodialysis
Brief Title: Results of Cold Stored Allografts in Vascular Access
Acronym: RAVASC
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI096
Record Dates: First submitted 2020-06-16; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: End Stage Renal Failure on Dialysis; Hemodialysis Access Failure
Keywords: Hemodialysis; Vascular access; Homologous vein; Allogenous vein graft; Cold stored venous allograft; Saphenous vein; Haemodialysis; Biological graft; Patency; Primary patency; Secondary patency; Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cold Stored Allograft Vascular Access
  Interventions: Procedure: Vascular access by pass using a cold stored venous allograft

INTERVENTIONS:
Procedure: Vascular access by pass using a cold stored venous allograft — Creation or surgical repair of a vascular access for hemodialysis using a cold venous allograft

SUMMARY:
Vascular access creation in patients with renal failure requiring long-term hemodialysis can be a challenge when there is no more autologous material or in case of infection, in a population undergoing long term dialysis with a longer life-expectancy. Many types of grafts have been used, with its advantages and drawbacks, such as prosthetic grafts (PTFE). Over the past decade, surgeons have used cold stored venous allografts as a biological conduit for hemodialysis, with the idea of avoiding most of major complications including a lower incidence of infection and steal syndrome, with patencies at least equivalent to PTFE. There is only a few data in the litterature, but many surgical teams use it when there is no autologous material or in case of infection.

The aim of the study is to give the primary patency of vascular access with this technique, and to assess its long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal failure patient requiring hemodialysis
* With the placement of a venous allograft for a hemodialysis approach
* Who underwent a surgery between January 1, 2014 and December 31, 2018 in a vascular surgery department participating in our study

Exclusion Criteria:

* Patient <18 years old, or under guardianship / curatorship
* Patient objecting to the use of his personal data in the context of research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patient with end-stage renal disease for whom a allograft was used for his hemodialysis access.
  * The patient can be treated on an ambulatory surgery or in full hospitalization
  * In the surgical departments having given their agreement to participate in our study
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Intervention free vascular access survival (in days) | 30 days
  The interval in days between the vascular access creation and the first successful re intervention (primary patency)
Intervention free vascular access survival (in days) | 6 months
  The interval in days between the vascular access creation and the first successful re intervention (primary patency)
Intervention free vascular access survival (in days) | 1 year
  The interval in days between the vascular access creation and the first successful re intervention (primary patency)
Intervention free vascular access survival (in days) | 2 years
  The interval in days between the vascular access creation and the first successful re intervention (primary patency)
Intervention free vascular access survival (in days) | 3 years
  The interval in days between the vascular access creation and the first successful re intervention (primary patency)

SECONDARY OUTCOMES:
Thrombosis free vascular access survival (in days) | 30 days
  The interval in days between the vascular access creation and the first occlusion with a successful re intervention (primary assisted pantency)
Thrombosis free vascular access survival (in days) | 90 days
  The interval in days between the vascular access creation and the first occlusion with a successful re intervention (primary assisted pantency)
Thrombosis free vascular access survival (in days) | 6 months
  The interval in days between the vascular access creation and the first occlusion with a successful re intervention (primary assisted pantency)
Thrombosis free vascular access survival (in days) | 1 year
  The interval in days between the vascular access creation and the first occlusion with a successful re intervention (primary assisted pantency)
Thrombosis free vascular access survival (in days) | 2 years
  The interval in days between the vascular access creation and the first occlusion with a successful re intervention (primary assisted pantency)
Thrombosis free vascular access survival (in days) | 3 years
  The interval in days between the vascular access creation and the first occlusion with a successful re intervention (primary assisted pantency)
Abandonment of the vascular access (in days) | 30 days
  The interval in days between the vascular access creation and its abandonment (secondary patency)
Abandonment of the vascular access (in days) | 90 days
  The interval in days between the vascular access creation and its abandonment (secondary patency)
Abandonment of the vascular access (in days) | 6 months
  The interval in days between the vascular access creation and its abandonment (secondary patency)
Abandonment of the vascular access (in days) | 1 year
  The interval in days between the vascular access creation and its abandonment (secondary patency)
Abandonment of the vascular access (in days) | 2 years
  The interval in days between the vascular access creation and its abandonment (secondary patency)
Abandonment of the vascular access (in days) | 3 years
  The interval in days between the vascular access creation and its abandonment (secondary patency)

OTHER OUTCOMES:
Early and late complications (in days) | 30 days
  The interval in days between the vascular access creation and the occurence of complications (stenosis, thrombosis, failure, hyperflow, distal ischemia, aneurysm)
Early and late complications (in days) | 90 days
  The interval in days between the vascular access creation and the occurence of complications (stenosis, thrombosis, failure, hyperflow, distal ischemia, aneurysm)
Early and late complications (in days) | 6 months
  The interval in days between the vascular access creation and the occurence of complications (stenosis, thrombosis, failure, hyperflow, distal ischemia, aneurysm)
Early and late complications (in days) | 1 year
  The interval in days between the vascular access creation and the occurence of complications (stenosis, thrombosis, failure, hyperflow, distal ischemia, aneurysm)
Early and late complications (in days) | 2 years
  The interval in days between the vascular access creation and the occurence of complications (stenosis, thrombosis, failure, hyperflow, distal ischemia, aneurysm)
Early and late complications (in days) | 3 years
  The interval in days between the vascular access creation and the occurence of complications (stenosis, thrombosis, failure, hyperflow, distal ischemia, aneurysm)
Incidence of the socio-demographic and clinical characteristics of the patients on secondary patency | 3 years
  Compare the duration of secondary patency according to the socio-demographic and clinical characteristics of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Vascular Surgery Nancy University Hospital, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidli J, Widmer MK, Basile C, de Donato G, Gallieni M, Gibbons CP, Haage P, Hamilton G, Hedin U, Kamper L, Lazarides MK, Lindsey B, Mestres G, Pegoraro M, Roy J, Setacci C, Shemesh D, Tordoir JHM, van Loon M, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Lindholt J, Naylor R, Vega de Ceniga M, Vermassen F, Verzini F, Esvs Guidelines Reviewers, Mohaupt M, Ricco JB, Roca-Tey R. Editor's Choice - Vascular Access: 2018 Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Jun;55(6):757-818. doi: 10.1016/j.ejvs.2018.02.001. Epub 2018 May 2. No abstract available. PMID 29730128
- [Background] Heintjes RJ, Eikelboom BC, Steijling JJ, van Reedt Dortland RW, van der Heijden FH, Bastini M, van der Graaf Y, Blankestijn PJ, Vos J. The results of denatured homologous vein grafts as conduits for secondary haemodialysis access surgery. Eur J Vasc Endovasc Surg. 1995 Jan;9(1):58-63. doi: 10.1016/s1078-5884(05)80226-6. PMID 7664014
- [Background] Schneider M, Barrou B, Cluzel P, Hamani A, Bitker MO, Richard F. [Value of preserved saphenous vein graft for the creation of access ports in hemodialyzed patients: report of 309 cases]. Prog Urol. 2003 Sep;13(4):585-91. French. PMID 14650287
- [Background] Berardinelli L. Grafts and graft materials as vascular substitutes for haemodialysis access construction. Eur J Vasc Endovasc Surg. 2006 Aug;32(2):203-11. doi: 10.1016/j.ejvs.2006.01.001. Epub 2006 Feb 20. PMID 16490368
- [Background] Nedved K, Suchy T, Halova J, Malicky M, Gorun P, Vitvar P. Allogenous vein graft as vascular access for hemodialysis--lost battle? J Vasc Access. 2012 Jul-Sep;13(3):366-73. doi: 10.5301/jva.5000062. PMID 22367646